CLINICAL TRIAL: NCT07321834
Title: A Phase 2, Randomized, Double-blind, Vehicle-Controlled, Multi-Center Clinical Trial Study to Evaluate Ready to Use Injectable AI-09 In Participants With Glabellar Lines
Brief Title: A Study to Evaluate AI-09 In Participants With Glabellar Lines
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eirion Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AI-09-GL-201
Record Dates: First submitted 2026-01-02; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Glabellar Lines
Keywords: Botulinum Toxin; Ready to use; Glabellar Lines; AI-09-GL-201

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Treatment (Experimental): AI-09
  Interventions: Biological: AI-09 Ready Use Injectable Botulinum Toxin
- Vehicle (Placebo Comparator): Vehicle
  Interventions: Biological: Vehicle

INTERVENTIONS:
Biological: AI-09 Ready Use Injectable Botulinum Toxin — AI-09 Ready Use Injectable Botulinum Toxin
  Arms: Active Treatment
Biological: Vehicle — Vehicle
  Arms: Vehicle

SUMMARY:
Phase 2 clinical study to evaluate the efficacy, safety, and tolerability of AI-09, a Ready-to-Use Liquid Injectable Botulinum Toxin.

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, out-patient, prospectively randomized, double-blind, vehicle-controlled, multi-center clinical study to evaluate the efficacy, safety, and tolerability of AI-09, a Ready-to-Use Liquid Injectable Botulinum Toxin, administered to participants with glabellar lines. The study is designed as a single dose study evaluating AI-09 at a dose of versus Vehicle.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 70 years of age
* moderate to severe glabellar lines (IGA 2 to 3) at maximum frown
* moderate to severe glabellar lines (SSA 2 to 3) at maximum frown
* willingness to refrain from the use of facial fillers, retinoids, Botox®, laser
* female participants of child-bearing potential must have a negative urine pregnancy test and be non-lactating at the Baseline (Day 0) visit and must utilize birth control throughout the study
* participants should be in good general health as determined by the investigator and free of any disease that may interfere with study evaluations or the Investigational Product

Exclusion Criteria:

* the inability to substantially lessen glabellar lines by physically spreading them apart
* eyelid ptosis, and/ or excessive weakness or atrophy in the target muscle(s)
* presence or history of "dry eye"
* history of periocular surgery, brow lift or related procedures, or deep dermal scarring
* concurrent or recent (within the last 6 months) use of any other botulinum toxin drug product anywhere in the body
* history of immunization or hypersensitivity to any botulinum toxin serotype
* history of non-response to any prior botulinum toxin treatments anticipated need for treatment with botulinum toxin of any serotype for any reason during the trial (other than the investigational treatment)
* any medical condition that may put the subject at increased risk with exposure to botulinum toxin including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other condition that might interfere with neuromuscular function
* pregnancy or lactation
* application of any topical prescription medication to the treatment area within 14 days prior to treatment
* participation in another investigational drug trial or receiving any investigational treatment(s) within 30 days of Baseline (Day 0)
* alcohol or drug abuse within the past 3 years
* refusal or inability with the subject's ability to give informed consent or comply with the requirements of the protocol for any reason

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2025-12-03 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
IGA-C | From enrollment (baseline) to the Week 04 Visit
  Change from Baseline (CfB) in IGA-C (Investigator Global Assessment on Contraction) as assessed using the 4-point Glabellar Line Severity Scale (GLS), with score "3" being Severe and score "0" being None.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Center for Clinical and Cosmetic Research, Aventura, Florida
  - Research Institute of the Southeast, Inc., West Palm Beach, Florida
  - Delricht Research, New Orleans, Louisiana
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Research Your Health, Plano, Texas

IPD SHARING:
Plan to Share IPD: No